CLINICAL TRIAL: NCT04373993
Title: Prehospital Minutes Count During a Stroke. Factors Associated With Prehospital Delays With Data From Various Regions in Norway and One Region in Switzerland
Brief Title: Prehospital Minutes Count During a Stroke.
Status: Active, not recruiting | Type: Observational
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/1729 REK
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-03

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Nordlandssykehuset HF
- Akershus universitetsssykehus
- Helgelandssykehuset
- Basel University Hospital

SUMMARY:
The ultimate objective is to improve the efficacy of prehospital procedures for patients suffering an acute stroke. Increased precision in prehospital selection and a more efficient transport chain will lead to an even more rapid start of treatment and thus benefit patients. The research project has two parts: one part collecting data from medical reports and one study with qualitative in-depth interviews. The project will gather data from various parts of Norway and from a University hospital in Switzerland for comparison between regions and countries. Data will be retrieved through intrahospital and prehospital medical records from various parts of Norway (Nordland Hospital, Akershus University Hospital and Helgeland Hospital) and from Basel University hospital in Switzerland. Knowledge of factors associated with delays will be compared for regions in the north and south of Norway, as well as abroad. The information obtained will be analysed to identify components in the chain that may be improved as concerns time saving.

ELIGIBILITY:
Inclusion Criteria:

• Final diagnosis of stroke at discharge from hospital

Exclusion Criteria:

• Hospital admission later than one week from stroke onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients discharged from the respective hospitals with a diagnosis of stroke during the period of inclusion.
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Time delay from ictus to hospital arrival | Within 4 hours
  Delay from first symptoms of stroke until arrival at hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Carlsson, Bodø, Norway